CLINICAL TRIAL: NCT05965999
Title: A Multicenter, Prospective, Open-Label Registry Study of the Utilization of EsoGuard, on Samples Collected Using EsoCheck, in an At-Risk Population Undergoing Standard of Care Screening for, and Management of, Previously Undiagnosed Barrett's Esophagus and/or Esophageal Adenocarcinoma
Brief Title: Lucid Registry Study
Acronym: Lucid Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Organization: PAVmed Inc. (Industry)
Other Study IDs: LUD-PR-0421
Record Dates: First submitted 2023-01-23; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Barretts Esophagus With Dysplasia; Barrett's Esophagus Without Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EsoCheck — EsoCheck® (EC) is an FDA 510(k) cleared device that is indicated for use in the collection and retrieval of surface cells of the esophagus in the general population 12 years of age and older.

SUMMARY:
This is a multicenter, prospective, observational study designed to capture a limited set of data consisting of diagnostic test results and clinical management information on subjects who undergo EC/EG to assess for the presence of BE/EAC. Once sufficient time has elapsed for EsoGuard results to be available, as well as for any subsequent clinical evaluation to have been performed (e.g., upper endoscopy and any initial therapeutic management), study staff will obtain the desired information and record it in an electronic data collection (EDC) system, pertaining to subject demographics, pertinent medical history, and risk factors for BE or EAC as well as (1) information about the EsoCheck cell collection procedure and patient tolerance, (2) EsoGuard test result; (3) initial clinical management including upper endoscopy, if performed, and diagnosis (as determined by the endoscopist and the pathologist assessing any biopsies taken), as well as (4) additional clinical management and/or a therapeutic procedure(s) performed. The time point for collecting such information shall be fluid, depending on the time course of care provided subsequent to the EsoGuard result being available. It is expected typically to be approximately 4 months given the systemic delays in scheduling and performing upper endoscopies and obtaining biopsy results. There is no a priori limit on the timeline for obtaining these data, but it is . anticipated that all data collection will be completed within 8 months of the availability of EsoGuard results.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females who have provided informed consent for prospective registry participation
2. Subject in whom the clinical decision has been made to screen for BE/EAC using EsoGuard testing on samples collected with EsoCheck

Exclusion Criteria:

1. Inability to provide written informed consent
2. Subjects who fall outside the eligible population defined by the EsoCheck device Instructions For Use (IFU)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have recently undergone or are scheduled to undergo EsoCheck administration (as prescribed by a licensed healthcare provider) will be invited to participate in the optional EsoGuard Registry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between positive EsoGuard test results and upper endoscopy diagnosis (i.e., subjects with BE/EAC newly diagnosed by upper endoscopy) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
The number of subjects with a positive EsoGuard test | Through study completion, an average of 1 year
Agreement between negative EsoGuard test results and upper endoscopy diagnosis (i.e., subjects determined not to have BE/EAC on upper endoscopy) | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gisella Lopez, Study Director — Lucid Diagnostics
Locations (1):
- LUCID DX, Lake Forest, California, United States

IPD SHARING:
Plan to Share IPD: No